CLINICAL TRIAL: NCT05995834
Title: Producing a Novel Symptom Burden Scale for People Living With Idiopathic Multicentric Castleman Disease (ISBUS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RECORDATI GROUP (Industry)
Collaborators: University of Sheffield (ScHARR) (Unknown); KMC Health Care (Unknown); Castleman Disease Collaborative Network (CDCN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ISBUS
Record Dates: First submitted 2023-07-26; First posted 2023-08-16 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Multicentric Castleman's Disease
MeSH Terms: conditions — Multi-centric Castleman's Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Research questions — Stage 1: Secondary analysis of a previous international survey to identify items
  Stage 2: Cognitive debriefing interviews with about 10 people living with iMCD to assess the content validity of the items
  Stage 3: Completion of questionnaire to finalise scale
  Stage 4a: Re-administering of follow-up questionnaire to Stage 3 patients to assess minimally important clinical difference. Test-retest will be calculated only in patients exhibiting no change.
  Stage 4b: Qualitative interviews with a subset of participants from Stages and 4 to help with interpretation of meaningful difference from their perspective

SUMMARY:
Development, validation of a novel symptom burden scale to assess and quantify the burden experienced by people living with Idiopathic Multicentric Castleman Disease (iMCD).

DETAILED DESCRIPTION:
Idiopathic Multicentric Castleman Disease (iMCD) is a rare lymphoproliferative disorder associated with systemic inflammation and organ dysfunction. The condition has an unknown aetiology and diagnostic criteria were established recently in 2017. It can be distinguished from other forms of Castleman Disease, including unicentric presentations and Multicentric Castleman Disease (MCD) that is associated with the Kaposi sarcoma herpesvirus. iMCD has an estimated prevalence of between 6.9 and 9.7 people per million. While clinical presentations vary, iMCD can be associated with a high degree of symptom burden, including constitutional, gastrointestinal, neuropsychiatric, dermatologic, respiratory, and hematologic or lymphoreticular problems. Both symptoms and the side-effects of treatment can impact the health-related quality of life (HRQoL) of people with iMCD

This international mixed-methods study will be conducted in four stages:

Stage 1: Item generation

* Drawing on the content, data, and analysis from a previous international patient online survey in iMCD with 65 patients, generate draft PROM content (including a longlist of candidate draft items under existing themes) to assess symptom burden in iMCD.
* Incorporate expert opinion and lived experience to achieve consensus on which items will be tested for inclusion in the symptom burden scale via an online multi-stakeholder workshop involving the funder, research team, patient and public involvement and engagement (PPIE) representative(s) (i.e., patients with iMCD and/or their carers), healthcare professionals, and any other relevant stakeholders.

Stage 2: Item testing and refinement

* Cognitive debriefing interviews with about 10 people living with iMCD to assess the content validity of the items (and associated PROM content) in terms of relevance, comprehensibility, and comprehensiveness. This will include assessing whether they are important/meaningful to patients.
* Analyse and summarise qualitative evidence on content validity, make recommendations on revisions to the draft PROM, and agree this with the multi-stakeholder advisory group (as described above) and a separate group of PPIE collaborators.

Stage 3: Final item selection

* Administer the refined PROM (from Stage 2) to as wide a sample as possible of people living with iMCD. The estimated sample size is 100 patients. The PROM will be administered alongside additional sociodemographic and clinical questions and measures of burden and/or health-related quality of life (HRQoL).
* Taking into account the sample size, conduct appropriate psychometric analyses in order to provide evidence for final item selection and to provide preliminary psychometric evidence on the reliability and validity of the final measure.
* Taking into account all of the available qualitative and quantitative evidence, and a consultation with PPIE collaborators, agree (with the multi-stakeholder advisory group) on final item selection, with the goal of obtaining an 8-10 item measure of symptom burden.

Stage 4: Preliminary measures of change

* Stage 4a: Re-administer the refined PROM (from Stage 2) to participants (from Stage 3) alongside measure(s) of perceived clinical change.
* Stage 4b: Conduct qualitative interviews with about 10 participants who have completed the PROM at both time points to understand what constitutes a meaningful difference from their perspective.
* Triangulate quantitative and qualitative data to estimate a minimally important clinical difference (MCID) for the new PROM, agreed with the multi-stakeholder advisory group.

Recruitment for Stages 2-4 will take place in USA, Canada, Brazil, Australia, New Zealand and the United Kingdom. Interviews will be conducted online for Stages 2 and 4 and the psychometric survey will be hosted and administered online.

Governance: The results of each stage will be discussed and final decisions will be made with a multi-stakeholder group consisting of the wider research team, clinicians and other healthcare professionals and PPIE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Multicentric Castleman Disease (iMCD)
* Adults (aged 18+ years)
* Fluent in English

Exclusion Criteria:

* No diagnosis of iMCD
* Children (aged < 18 years)
* Not able to understand or communicate in English
* People lacking the capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with idiopathic Multicentric Castleman Disease (iMCD).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Long list of candidate items for the scale (stage 1) | Sept 2023 - Nov 2023
  completion of data analysis from a previous survey
Completion of interviews (stage 2) | Within 6 months from start (With this being a rare condition, data from all patients will be collected at various levels of treatment and time from diagnosis)
  completion of interviews by 10 patients from all recruiting sites
Completion of questionnaire (stage 3) | Within 9 months from start (With this being a rare condition, data from all patients will be collected at various levels of treatment and time from diagnosis). NB: Advisory comments noted.
  completion of questionnaire which includes extra questions about treatments, time of diagnosis.
  Completion of EQ-5D for external validity of PROM. NB: EQ-5D is the full name of the instrument and not an acronym.
Completion of follow-up questionnaire (stage 4a) | About 8 weeks after Stage 3 questionnaire. Note: Advisory comments noted.
  completion of follow-up questionnaire from Stage 3 by same patients who participated in Stage 3. Note: The full name of the scale will be discussed and confirmed. At the moment, the working title is Idiopathic Multicentric Castleman Disease Symptom Burden Scale (ISBUS).
Completion of interviews (stage 4b) | About 4 weeks after Stage 4a
  completion of interviews by 10 patients from all recruiting sites

CONTACTS AND LOCATIONS:
Overall Officials: Anju Keetharuth, PhD, Principal Investigator — University of Sheffield; Philip Powell, PhD, Principal Investigator — University of Sheffield

IPD SHARING:
Plan to Share IPD: No
Deanonymized transcriptions of stages 2 and 4 interviews will be securely stored in the University of Sheffield repository with access restricted to investigators only. Quantitative data from stages 3 and 4a will be processed, stored and accessed similarly in the same location.

REFERENCES:
- See also: example of registration of PROMs — https://clinicaltrials.gov/study/NCT03052283?term=Development%20PROM&rank=3
- See also: example of registration of PROMs — https://clinicaltrials.gov/study/NCT05274867?term=Development%20PROM&rank=6
- See also: example of registration of PROMs — https://clinicaltrials.gov/study/NCT05315765?term=Development%20PROM&rank=8